CLINICAL TRIAL: NCT03493503
Title: Efficacy of a Loading Dose of IV Salbutamol in Children Admitted to a PICU for Severe Acute Asthma or Severe Acute Wheeze
Brief Title: Status Asthmaticus on the PICU; Intravenous Salbutamol
Acronym: STATIC IV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Matthijs de Hoog, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL55029.078.16
Record Dates: First submitted 2018-03-12; First posted 2018-04-10 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Childhood Asthma With Status Asthmaticus
MeSH Terms: interventions — Albuterol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Salbutamol loading dose (Experimental): Salbutamol loading dose of 15 mcg/kg in 10 minutes, with a maximum of 750 mcg.
  Interventions: Drug: Salbutamol
- Sodium Chloride 0.9% (Placebo Comparator): 10 ml of Sodium Chloride 0.9% in 10 minutes.
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Salbutamol — Intravenous Salbutamol loading dose
  Arms: Salbutamol loading dose
Drug: Sodium Chloride 0.9% — 10 ml of Sodium Chloride 0.9% in 10 minutes intravenous
  Arms: Sodium Chloride 0.9%

SUMMARY:
Although IV salbutamol is frequently used in children in a wide range, pharmacodynamic data are scarce. To date, there is an insufficient evidence base to guide initial and subsequent dosing recommendation for its IV use in children. Especially the need for a loading dose needs to be addressed. Therefore, pharmacodynamic and kinetic data are needed to guide initial dosing strategies of IV salbutamol in children. To assess the efficacy of a loading dose of intravenous salbutamol in children admitted to a PICU for severe acute wheeze or severe acute asthma. Efficacy is measured by the reduction in asthma score (Qureshi) at 1 hour after administration of the loading dose, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Between 2-18 years of age at moment of inclusion
* Admitted to PICU for Severe Acute Asthma or Severe acute (viral) wheeze
* Requiring administration of IV salbutamol

Exclusion Criteria:

* Patient is outside of specified age range
* Patient has already received a -loading dose- of IV salbutamol in the general hospital
* Lower airway infection with consolidation on a chest X ray -Patient has Down's Syndrome
* Patient has a congenital/acquired heart defect that interferes with normal asthma treatment
* Patient has a primary/secondary immunodeficiency
* Patient has a pre-existing chronic pulmonary condition, known to mimic asthma: Cystic fibrosis, Bronchopulmonary dysplasia, Bronchiolitis obliterans

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
Reduction Asthma score | First 24 hours after admission on the PICU
  The primary outcome variable is (reduction of) asthma score (Qureshi) 1 hour after administration of loading dose in the intervention group compared to the placebo group. Based on expert opinion, we consider a reduction of 2 points to represent a clinically relevant improvement.

SECONDARY OUTCOMES:
Cumulative dose of IV salbutamol | Through study completion, an average 48 hours
Maximum infusion rate of IV salbutamol in mcg/kg/min | Through study completion, an average 48 hours
Total duration of IV salbutamol treatment in hours | Through study completion, an average 48 hours
Occurrence/frequency of side effects | Through study completion, an average 48 hours
Length of Stay on PICU in days | Through study completion, an average 72 hours
Use of co-medication | Through study completion, an average 72 hours
Use of/duration of non-invasive mechanical ventilation in days | Through study completion, an average 72 hours
DNA polymorphism of the ADRB2-receptor gene | Through study completion, an average 1 year
  The investigators will look at DNA, if there is a polymorphism in the ADRB2-receptor gene. If there is a polymorphism it can cause downregulation of the adrenergic B2 receptors.
Use of/duration of non-invasive/invasive mechanical ventilation in days | Through study completion, an average 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands